CLINICAL TRIAL: NCT01535989
Title: A Phase I Study of Inotuzumab Ozogamicin (CMC-544) in Combination With Temsirolimus (CCI-779) in Patients With Relapsed or Refractory CD22-positive B-cell Non Hodgkin's Lymphomas
Brief Title: Study of Inotuzumab Ozogamicin + Temsirolimus in Patients With Relapsed or Refractory CD22+ B-cell NHLymphoma
Acronym: IOSI-LND-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cristiana Sessa (Other)
Responsible Party: Sponsor-Investigator, Cristiana Sessa, Prof., Oncology Institute of Southern Switzerland
Organization: Oncology Institute of Southern Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOSI-LND-001
Record Dates: First submitted 2012-01-27; First posted 2012-02-20 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: B-cell Lymphoma Refractory
Keywords: B-cell Non Hodgkin's Lymphomas; CD22 positive
MeSH Terms: interventions — Inotuzumab Ozogamicin; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intravenous (Experimental): dose escalation
  Interventions: Drug: Inotuzumab Ozogamicin; Drug: Temsirolimus

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — starting dose 0.8 mg/m2, d1 administration, q4wks
  Other Names: CMC-544
Drug: Temsirolimus — starting dose of 15mg, weekly administration, q4ws
  Other Names: Torisel, CCI-779

SUMMARY:
This is an open label phase I study of Inotuzumab Ozogamicin, an antibody-targeted intravenous chemotherapy agent composed of a CD22-targeted antibody linked to calicheamicin, in combination with the mammalian target of rapamycin (mTOR) inhibitor Temsirolimus, in patients with relapsed/refractory CD22+ B-cell non Hodgkin's lymphomas (NHLs). Both Inotuzumab Ozogamicin and Temsirolimus have been evaluated as single agents as well as in combination with rituximab in patients with NHLs. This is the first study combining the two agents together. In the present study Inotuzumab Ozogamicin will be administered intravenously on d1 at the starting dose of 0.8 /m2. Temsirolimus will be administered intravenously on days 1,8,15 and 22 at the starting dose of 15mg. Cycles will be repeated every 28 days.

ELIGIBILITY:
Key inclusion criteria

* Histologically and/or cytologically confirmed relapsed or refractory CD22+ B-cell Non Hodgkin's Lymphomas
* No limitations on prior treatments. Patients must have progressed after at least one prior therapy.
* Adult patients (aged > 18yrs old).
* ECOG status ≤ 1.
* Life expectancy greater than 3 months.
* Adequate organ and marrow function.

Key exclusion criteria

* Uncontrolled intercurrent illness
* Chronic obstructive or chronic restrictive pulmonary disease
* Hepatitis B, C and HIV
* Patients with known known central nervous system lymphoma involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
number of participants with adverse events based on the CTCAE v.4 | toxicities will be assessed during the participation of each patient in the study, an expected average of 8 weeks
  To determine the safety profile, establish the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of Inotuzumab Ozogamicin in combination with Temsirolimus in patients with relapsed/refractory CD22+ B-cell NHLs

SECONDARY OUTCOMES:
Antitumor activity based on Cheson criteria | after 12-18 months form the first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Stathis, Dr., Principal Investigator — Oncology Institute of Southern Switzerland
Locations (3):
- Switzerland (3):
  - InselSpital, Universitätsspital Bern, Bern, Canton of Bern
  - Oncology Institute of Southern Switzerland, Bellinzona, Canton Ticino
  - Kantonsspital St.Gallen, San Gallen, San Gallen

REFERENCES:
- [Derived] Pirosa MC, Zhang L, Hitz F, Novak U, Hess D, Terrot T, Pascale M, Mazzucchelli L, Bertoni F, Cavalli F, Zucca E, Stathis A. A phase I trial of inotuzumab ozogamicin in combination with temsirolimus in patients with relapsed or refractory CD22-positive B-cell non-Hodgkin lymphomas. Leuk Lymphoma. 2022 Jan;63(1):117-123. doi: 10.1080/10428194.2021.1966780. Epub 2021 Aug 19. PMID 34407735